CLINICAL TRIAL: NCT01396057
Title: A 6-month Multicenter, Randomized, Double-masked Phase IIIb-study Comparing the Efficacy and Safety of Ranibizumab Intravitreal Injections Versus Dexamethasone Intravitreal Implant in Patients With Visual Impairment Due to Macular Edema Following Branch Retinal Vein Occlusion (BRVO)
Brief Title: Efficacy and Safety of Ranibizumab Intravitreal Injections Versus Dexamethasone Intravitreal Implant in Patients With Branch Retinal Vein Occlusion (BRVO)
Acronym: COMRADE-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002EDE17; 2011-001019-30 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Visual Impairment; Macular Edema; Branch Retinal Vein Occlusion
Keywords: Visual impairment; macular edema; branch retinal vein occlusion; Dexamethasone implant; Ranibizumab
MeSH Terms: conditions — Vision Disorders; Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab; Dexamethasone; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ranibizumab (Experimental): Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitreally
  Interventions: Drug: Ranibizumab
- Dexamethasone (Sham Comparator): Intravitreal implant as per commercial label (700 μg Dexamethasone; long acting release (LAR) over 6 months
  Interventions: Other: Dexamethasone Implant; Other: Sham injection

INTERVENTIONS:
Drug: Ranibizumab — Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitreally. Ranibizumab was formulated as a sterile solution aseptically filled in a sterile glass vial. It was suitable for single use only and the content of the vial was not allowed to be split
  Arms: Ranibizumab
Other: Dexamethasone Implant — Comparator Ozurdex® (dexamethasone) was formulated as a rod shaped implant to be inserted into the eye by an applicator. The implant as well as the respective applicator were suitable for single use only.
  Arms: Dexamethasone
Other: Sham injection — Sham injection: Empty sterile syringes were provided so that masking could be maintained. Either empty syringes in the case of sham injections or pre-filled syringes in the case of ranibizumab injections were visible to the patient in the room of study drug administration
  Arms: Dexamethasone

SUMMARY:
This clinical trial is designed to compare ranibizumab in comparison with Dexamethasone implant after 6 months of treatment. In the study arm Ranibizumab will be given monthly in a pro re nata scheme whereas the comparator Dexamethasone implant is given once at Month 0 with sham injections PRN afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with visual impairment due to macular edema following BRVO
* Diagnosis of BRVO at maximum 6 months prior to Screening
* BCVA using ETDRS charts of 20/40 to 20/400 in the study eye

Exclusion Criteria:

* Media clarity, pupillary dilation and patient cooperation not sufficient for adequate fundus photographs
* Central retinal thickness (CRT) < 250 µm in the study eye
* Prior episode of RVO in the study eye
* Active formation of new vessels in the study eye
* Anti-VEGF-treatment in the study or the fellow eye 3 months prior to Baseline
* IOP ≥ 30mmHg or uncontrolled glaucoma; patients may be re-screened after 1 month if they have undergone glaucoma treatment
* Improvement of > 10 letters on BCVA between Screening and Baseline

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- Novartis Investigative Site, Prague, Czechia
- Germany (37):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Regensburg, Germany
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Rothenfelde
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg I. Br
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Ingolstadt
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Sulzbach
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würzburg
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Poland (2):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bytom
- United Kingdom (17):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Derby
  - Novartis Investigative Site, Gloucester
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Rugby
  - Novartis Investigative Site, Westcliff-on-Sea
  - Novartis Investigative Site, York

REFERENCES:
- [Derived] Shalchi Z, Mahroo O, Bunce C, Mitry D. Anti-vascular endothelial growth factor for macular oedema secondary to branch retinal vein occlusion. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD009510. doi: 10.1002/14651858.CD009510.pub3. PMID 32633861

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab | Dexamethasone
Started | 126 | 118
Completed | 115 | 100
Not Completed | 11 | 18
Not completed — Adverse Event | 2 | 6
Not completed — Unsatisfactory therapeutic effect | 2 | 6
Not completed — Protocol deviation | 4 | 4
Not completed — Consent withdrawn | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Dexamethasone | Total
Number analyzed (Participants) | 126 | 118 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (10.9) | 65.6 (10.0) | 65.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 57 | 133
  Male | 50 | 61 | 111

OUTCOME MEASURES:

1. Primary Outcome: Mean Average Best Corrected Visual Acuity (BCVA) Change From Month 1 Through Month 6 to Baseline
Description: the average of the changes in BCVA (letters) from baseline to any post-baseline visit, i.e. the mean of six differences to baseline for the six post-baseline visits at month 1 to 6
Time Frame: Baseline, month 6
Population: The Full Analysis Set (FAS) consisted of all patients from the Randomized Set (RS) who had received at least one application of study treatment and had at least one post-baseline assessment for BCVA. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Letters | 14.9 (9.9) | 10.1 (9.5)

2. Secondary Outcome: Mean BCVA Change From Baseline to Endpoints Month 1 to Month 6
Description: The analysis was performed by an analysis of covariance (ANCOVA) model with average change in BCVA (letters) from Visit 1 through Visit 6 as dependent variable, and with the factors center, treatment and covariate baseline BCVA as predictors
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Letters (EDTRS)
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Letters (EDTRS) | 16.18 [14.04 to 18.32] | 8.10 [5.79 to 10.40]

3. Secondary Outcome: Percentage of Patients Gaining / Losing ≥ 15 / 10 / 5 Letters After 6 Month Treatment
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who gained 15, 10 or 5 more letters of visual acuity at month 6 as compared with baseline
Time Frame: Baseline, 6 month
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Participants
  Gain≥15 letters | 77 | 44
  Loss of ≥15 letters | 0 | 6
  Gain ≥10 letters | 97 | 63
  Loss of ≥10 letters | 2 | 8
  Gain ≥5 letters | 108 | 76
  Loss of ≥5 letters | 4 | 14

4. Secondary Outcome: Time to Achieve a Significant Improvement ≥ 15 Letters
Description: The time was analyzed by the Kaplan-Maier-Method, adjusting the calculation for dropouts
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Time to event (Days)
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Time to event (Days) | 63 [56 to 84] | 64 [59 to 126]

5. Secondary Outcome: Change Over Time in BCVA
Description: as for outcome 2
Time Frame: baseline, month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Letters
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Letters
  Month 1 | 10.35 [8.53 to 12.17] | 10.44 [8.48 to 12.40]
  Month 2 | 13.84 [12.04 to 15.64] | 12.62 [10.69 to 14.56]
  Month 3 | 15.52 [13.44 to 17.59] | 9.16 [6.92 to 11.39]
  Month 4 | 14.39 [12.38 to 16.41] | 8.59 [6.42 to 10.76]
  Month 5 | 14.65 [12.52 to 16.78] | 9.08 [6.79 to 11.37]
  Month 6 | 16.18 [14.04 to 18.32] | 8.10 [5.79 to 10.40]

6. Secondary Outcome: Change Over Time of the Central Retinal Thickness (CRT)
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT). The images were reviewed by a central reading center to ensure a standardized evaluation
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
µm | -230.6 (169.3) | -112.3 (172.1)

7. Secondary Outcome: Changes in the Quality of Life According to the National Eye Institute Visual Function Questionnaire (NEI-VFQ 25) Questionnaires
Description: The VFQ-25 composite and subscale scores range from 0 to 100, a higher score indicating better functioning. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated improvement in quality of life due to vision function.
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Score on a scale | 7.2 (10.2) | 2.8 (12.6)

8. Secondary Outcome: Changes in the Quality of Life According to the Short Form (36) Health Survey (SF-36)Questionnaires
Description: SF-36 summary measures are norm-based scores with mean = 50 and SD = 10. Higher scores indicate better health
Time Frame: Baseline, month 6
Population: The Full Analysis Set (FAS) consisted of all patients from the Randomized Set (RS) who had received at least one application of study treatment and had at least one post-baseline assessment for BCVA. observed is only described in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Units on a scale
  SF-36 physical component (n=121,114) | -1.1 (5.7) | -0.4 (5.7)
  SF-36 mental component (n=121,114) | 3.3 (9.2) | 0.2 (9.6)

9. Secondary Outcome: Changes in the Quality of Life According to Euro Quality of Life (EQ-5D) Questionnaires
Description: The EQ-5D visual analog scale ranges from 0 to 100, 0 representing the worst and 100 the best imaginable health state.
Time Frame: Baseline, month 6
Population: The Full Analysis Set (FAS) consisted of all patients from the Randomized Set (RS) who had received at least one application of study treatment and had at least one post-baseline assessment for BCVA. Observed participants are only described in this analysis
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 123 | 118
Units on a scale | 0.7 (15.2) | -2.4 (15.4)

10. Secondary Outcome: Rate of the Internal Ocular Pressure (IOP)
Description: The proportion of patients with ≥ 10% increase in IOP compared to baseline at any post-baseline visit.
Time Frame: Baseline, month 6
Population: The Safety Set consisted of all patients from the RS who had received at least one application of study treatment and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received. The statement that a patient had no adverse events also constituted a safety assessment
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 126 | 118
Participants | 79 | 106

ADVERSE EVENTS:
Arm/Group | Ranibizumab | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 7/126 | 9/118
Other Adverse Events (participants affected / at risk) | 71/126 | 89/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=126) | Dexamethasone (N=118)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
BRADYARRHYTHMIA (Cardiac disorders) | 1 | 0
CONJUNCTIVITIS (Study eye) (Eye disorders) | 0 | 1
OCULAR HYPERTENSION (Study eye) (Eye disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1
FATIGUE (General disorders) | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
CELLULITIS (Study eye) (Infections and infestations) | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
KIDNEY RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
PERIRENAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1
SPLENIC INJURY (Injury, poisoning and procedural complications) | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
RHEUMATIC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
URETHRAL PROLAPSE (Renal and urinary disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=126) | Dexamethasone (N=118)
ABNORMAL SENSATION IN EYE (Study eye) (Eye disorders) | 5 | 3
BLEPHARITIS (Fellow eye) (Eye disorders) | 1 | 3
BLEPHARITIS (Study eye) (Eye disorders) | 2 | 5
CATARACT (Study eye) (Eye disorders) | 1 | 4
CONJUNCTIVAL HAEMORRHAGE (Study eye) (Eye disorders) | 12 | 14
CONJUNCTIVAL IRRITATION (Study eye) (Eye disorders) | 4 | 4
CONJUNCTIVITIS (Study eye) (Eye disorders) | 4 | 2
EYE DISCHARGE (Study eye) (Eye disorders) | 5 | 5
EYE IRRITATION (Fellow eye) (Eye disorders) | 1 | 3
EYE IRRITATION (Study eye) (Eye disorders) | 3 | 6
EYE PAIN (Study eye) (Eye disorders) | 9 | 13
EYELID OEDEMA (Study eye) (Eye disorders) | 0 | 3
FOREIGN BODY SENSATION IN EYES (Study eye) (Eye disorders) | 8 | 4
GLAUCOMA (Study eye) (Eye disorders) | 1 | 3
LACRIMATION INCREASED (Fellow eye) (Eye disorders) | 2 | 4
LACRIMATION INCREASED (Study eye) (Eye disorders) | 7 | 4
MACULAR OEDEMA (Study eye) (Eye disorders) | 4 | 7
OCULAR DISCOMFORT (Study eye) (Eye disorders) | 2 | 8
OCULAR HYPERAEMIA (Study eye) (Eye disorders) | 16 | 21
OCULAR HYPERTENSION (Study eye) (Eye disorders) | 0 | 6
RETINAL EXUDATES (Study eye) (Eye disorders) | 7 | 3
VISION BLURRED (Study eye) (Eye disorders) | 6 | 2
VISUAL ACUITY REDUCED (Study eye) (Eye disorders) | 4 | 6
VITREOUS DETACHMENT (Study eye) (Eye disorders) | 3 | 7
VITREOUS FLOATERS (Study eye) (Eye disorders) | 3 | 3
VOMITING (Gastrointestinal disorders) | 0 | 3
CYSTITIS (Infections and infestations) | 4 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 4
NASOPHARYNGITIS (Infections and infestations) | 20 | 21
FALL (Injury, poisoning and procedural complications) | 6 | 3
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 4
INTRAOCULAR PRESSURE INCREASED (Investigations) | 3 | 19
INTRAOCULAR PRESSURE INCREASED (Study eye) (Investigations) | 2 | 17
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 1
HEADACHE (Nervous system disorders) | 13 | 11
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 3
HYPERTENSION (Vascular disorders) | 7 | 5
VASCULAR SHUNT (Study eye) (Vascular disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety